CLINICAL TRIAL: NCT07049198
Title: The Effect of a Real-time 2D Motion Capture and Visual Feedback Gait Training Systems on Walking Performance in People With Unilateral Transfemoral Amputation
Brief Title: Real-time Motion Capture and Visual Feedback for Amputation Gait Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Hui-Ting Shih, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYCU114067AE
Record Dates: First submitted 2025-05-13; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Unilateral Transfemoral Amputation; Unilateral Knee Disarticulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time 2D motion capture and visual feedback system gait training group (VF) (Experimental): The VF group, the 2D motion capture and visual feedback training group, received an intervention consisting of 10 minutes of strength training followed by 30 minutes of visual feedback gait training using the 2DMV system.
  Interventions: Device: Real-time 2D motion capture and visual feedback system gait training
- Conventional physical therapy group (PT) (Active Comparator): The PT group, the conventional physical therapy group, received an intervention consisting of 10 minutes of strength training followed by 30 minutes of gait training without the use of the 2DMV system for visual feedback. During gait training, the therapist provided standard gait correction feedback typically used in conventional physical therapy.
  Interventions: Other: Conventional physical therapy group

INTERVENTIONS:
Device: Real-time 2D motion capture and visual feedback system gait training — The difference between the VF group and the PT group lies in the use of real-time visual feedback during gait training; the VF group receives real-time visual feedback, while the PT group undergoes gait training without visual feedback.
  Arms: Real-time 2D motion capture and visual feedback system gait training group (VF)
Other: Conventional physical therapy group — Ten minutes of strength training followed by thirty minutes of gait training, during which the 2DMV system is not used to provide visual feedback. During the gait training, the therapist provides gait correction feedback typically used in conventional physical therapy.
  Arms: Conventional physical therapy group (PT)

SUMMARY:
People with transfemoral amputation face challenges such as gait asymmetry, instability, and increased energy consumption due to loss of the knee joint. Because of the loss of proprioceptive feedback from their missing limbs, visual feedback is essential for gait correction. Additionally, current visual feedback systems lack portability, cost-effectiveness, and they fail to provide precise, intuitive feedback on spatiotemporal parameters, joint angles, and both frontal and sagittal plane information, limiting their effectiveness in correcting gait abnormalities.This study aims to investigate whether gait training using a real-time 2D motion capture and visual feedback gait training system (2DMV) can improve the gait biomechanics and psychosocial functions of people with unilateral transfemoral amputation (uTFA). The 2DMV system analyzes spatiotemporal parameters and joint kinematics during gait and displays the uTFA's image on a screen, providing visual feedback specifically targeting gait abnormalities. This allows individuals with uTFA to intuitively understand the feedback and make real-time gait adjustments. The biomechanical parameters include joint kinematics, gait symmetry, and walking performance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Individuals with unilateral transfemoral amputation or knee disarticulation
* Wear a prosthesis for at least 3 hours per day
* Have been using a prosthesis for more than 6 months
* Medicare Functional Classification Level (K-level) of 2 or above
* Able to walk independently for 5 meters without assistive devices
* No pain caused by poor prosthetic fit
* Montreal Cognitive Assessment Taiwan Version (MoCA-T) score ≥ 26

Exclusion Criteria:

* Uncontrolled systemic diseases (e.g., diabetes mellitus, hypertension)
* Cardiopulmonary or cardiovascular diseases (e.g., heart failure, severe asthma)
* History of neurological conditions that affect movement (e.g., stroke, spinal cord injury, cerebellar injury)
* Vestibular disorders
* Severe osteoporosis
* Other musculoskeletal injuries or open wounds
* Epilepsy
* Uncorrected visual impairments
* Congenital limb deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Step width ratio | The step width ratio will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  Step width ratio is calculated by dividing step width by pelvis width (step width/pelvis width), and the normal range is between 0.4 to 1.1.
Step length ratio | The step length ratio will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  Step length ratio is calculated by dividing the step length of the amputated limb by the step length of the non-amputated limb (a value closer to 1 indicate more symmetry, the step length of amputated limb is calculated as the distance between the heel of the non-amputated limb when initial contact and the heel of the amputated limb when initial contact; the step length of non-amputated limb is calculated as the distance between the heel of the amputated limb when initial contact and the heel of the non-amputated limb when initial contact)
Stride time ratio | The stride time ratio will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  Stride time ratio is calculated by dividing the stride time of the amputated limb by the stride time of the non-amputated limb (a value closer to 1 indicates more symmetry, the stride time of the amputated limb is calculated as the time from initial contact of the amputated limb to next initial contact of the same limb; the stride time of the non-amputated limb is calculated as the time from initial contact of the non-amputated limb to next initial contact of the same limb).
Stance time ratio | The stance time ratio will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  Stance time ratio is calculated by dividing the stance time of the amputated limb by the stance time of the non-amputated limb (a value closer to 1 indicates more symmetry, the stance time is calculated from initial contact to toe off of the same limb).
Swing time ratio | The swing time ratio will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  Swing time ratio is calculated by dividing the swing time of the amputated limb by the swing time of the non-amputated limb (a value closer to 1 indicates more symmetry, the swing time is calculated from toe off to initial contact of the same limb).
Hip extension angle | The hip extension angle will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The hip extension angle is measured in the sagittal plane during terminal stance.
Hip flexion angle | The hip flexion angle will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The hip flexion angle is measured in the sagittal plane at the maximum angle of hip flexion during the swing phase.
Trunk extension and flexion angle | The trunk extension and flexion angle will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The trunk extension and flexion angle is measured in the sagittal plane at the initial contact and terminal stance.
Hip adduction and abduction angle | The hip adduction and abduction angle will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The hip adduction and abduction angle is measured in the coronal plane at the maximum angle of hip adduction or abduction angle during the swing phase.
Horizontal pelvis tilt angle | The horizontal pelvis tilt angle will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The horizontal pelvis tilt angle is measured in the coronal plane at the maximum pelvis tilt angle during single-leg stance.
Trunk lateral flexion angle | The trunk lateral flexion angle will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The trunk lateral flexion angle is measured in the coronal plane during midstance.

SECONDARY OUTCOMES:
The Component Timed-Up-and-Go test, cTUG | The Component Timed-Up-and-Go test will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The participant will first be instructed to sit on a chair with a backrest. When the assessor says 'go,' the participant will stand up, walk forward, circle around a cone, return to the chair, and sit down, all at a self-selected speed. The assessor will time the duration of the entire process. The timing of the Component Timed-Up-and-Go test will be divided into five components: standing up, walking forward, circling around the cone, walking back to the chair, and sitting down. Time will be measured in seconds.
Gait speed | The gait speed will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  Gait speed will be measured by the assessor with a timer. The participant will be instructed to walk 5 meters at a self-selected speed. The first and last 1 meter will serve as the acceleration and deceleration phases, while the gait speed in middle 3 meters will be measured. Time will be measured in seconds.
The Activities-specific Balance Confidence Scale, ABC scale | The Activities-specific Balance Confidence Scale will be measured at Day 1, before the 1st intervention session, and after the 12th intervention session.
  The Activities-specific Balance Confidence Scale is a self-reported questionnaire used to assess balance confidence. Scores range from 0% to 100%, with higher scores indicating greater confidence. The scale consists of 16 items in total.
The National Aeronautics and Space Administration Task Load Index, NASA-TLX | The National Aeronautics and Space Administration Task Load Index will be measured after the 12th intervention session.
  The National Aeronautics and Space Administration Task Load Index is a self-repoted scale, totally has 6 items, including mental demand, physical demand, temporal demand, performance, effort, and frustration. The score will recorded as 0 to 100, with the higher score indicating higher work load.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

REFERENCES:
- See also: Related Info — https://iloveneuro.wixsite.com/ym-neuropt-lab-eng